CLINICAL TRIAL: NCT01290276
Title: Phase Ia/Ib Study of Normal Healthy Volunteer Clinical Trial of a Novel Ondansetron Formulation
Brief Title: Open-label, Normal Healthy Volunteer Clinical Trial of a Novel Ondansetron Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tong Lee (Other)
Responsible Party: Sponsor-Investigator, Tong Lee, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00024378; 110034 (Pro00024378) (Other: FDA IND); 110195 (Pro00026674) (Other: FDA IND); Pro00026674
Record Dates: First submitted 2011-01-09; First posted 2011-02-04 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Ondansetron; Methylphenidate
MeSH Terms: interventions — Ondansetron; Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ond-PR1 followed by (Ond-PR1 + MPh-IR) (Experimental): Oral dose of 8 mg of ondansetron pulsatile-release formulation 1 followed by Oral dose of 8 mg of ondansetron pulsatile-release formulation 1 (Ond-PR1) plus 10 mg methylphenidate immediate release (Mph-IR)
  Interventions: Drug: Ond-PR1; Drug: Ond-PR1 + MPh-IR; Drug: Ond-PR2; Drug: Ond-PR2 +_ MPh-IR
- Ond-PR2 followed by (Ond-PR2 + MPh-IR) (Experimental): Oral dose of 8 mg of ondansetron pulsatile-release formulation 2 followed by Oral dose of 8 mg of ondansetron pulsatile-release formulation 2 (Ond-PR2) plus 10 mg methylphenidate immediate release (Mph-IR)
  Interventions: Drug: Ond-PR1; Drug: Ond-PR1 + MPh-IR; Drug: Ond-PR2; Drug: Ond-PR2 +_ MPh-IR

INTERVENTIONS:
Drug: Ond-PR1 — Single oral dose of 8 mg of ondansetron pulsatile-release formulation 1 (Ond-PR1)
  Other Names: Zofran (ondansetron hydrochloride)
Drug: Ond-PR1 + MPh-IR — Single oral dose of 8 mg of ondansetron pulsatile-release formulation 1 (Ond-PR1) plus 10 mg methylphenidate immediate release (Mph-IR)
  Other Names: Zofran (ondansetron hydrochloride); Ritalin (methylphenidate hydrochloride)
Drug: Ond-PR2 — Single oral dose of 8 mg ondansetron pulsatile-release formulation 2 (Ond-PR2)
  Other Names: Zofran (ondansetron hydrochloride)
Drug: Ond-PR2 +_ MPh-IR — Single oral dose of 8 mg of ondansetron pulsatile-release formulation 2 (Ond-PR2) plus 10 mg methylphenidate immediate release (Mph-IR)
  Other Names: Zofran (ondansetron hydrochloride); Ritalin (methylphenidate hydrochloride)

SUMMARY:
The goals of this open-label Phase Ia study are to evaluate the Pharmacokinetics (PK) profiles of new novel single-dose Ondansetron Pulsatile Release (Ond-PR) formulations in normal healthy volunteers. After this initial phase, the investigators will follow with the Phase Ib study to determine Pharmacokinetic/Pharmacodynamic (PK/PD), safety, and tolerability interactions following simultaneous administration of these ondansetron formulations with a 10 mg Methylphenidate Immediate Release (MPh-IR) tablet in normal healthy volunteers.

DETAILED DESCRIPTION:
We will compare 2 different pulsatile-release formulations of ondansetron, PR1 and PR2. Ond-PR1 is a pH-sensitive formulation while Ond-PR2 is osmotic-sensitive.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent to participate in the study prior to screening. Consent will be documented by the subject's dated signature that will be counter-signed and dated by a witness.
* Healthy non-smoking, by history, adult male and/or female volunteers between the ages of 18 and 45 years old and with a Body Mass Index (BMI) of ≥18-≤32 kg/m2.
* Subjects must be in good health as determined by screening medical history, physical examination, vital signs, electrocardiogram, blood chemistry, hematology, and urinalysis (U/A) performed at screening.
* Normal Hematology Clinical Laboratory, Results, including: Normal White Blood Cell (WBC) and differential, Hematocrit, Hemoglobin, Platelet Counts
* Normal Electrocardiogram (ECG) and a measure between Q wave and T wave in the heart's electrical cycle at baseline (QTcB) ≤ 430 msec (males) or ≤ 430 msec (females)

Exclusion Criteria:

* Male and/or female subjects who consume more than 28 units of alcohol per week (one unit of alcohol equals ½ pint of beer, 4 ounces of wine, or 1 ounce of spirits) or those subjects who have a significant history of alcoholism or drug/chemical abuse within the last 2 years. Subjects must agree to abstain from alcohol, cola, tea, coffee, chocolate and other caffeinated drink and food from 2 days before Period 1, Day 1 and throughout confinement.
* Subjects who have used tobacco products or nicotine-containing products (including smoking cessation aids, such as gums or patches) within 3 months prior to Day -1.
* Subjects with positive results on tests for drugs of abuse, or alcohol at screening and check-in.
* Concomitant Medications: Any drugs, vitamins, over the counter (OTC) medicines and nutraceuticals if used within the previous 7 days of check-in as deemed clinically significant by the Principal Investigator (PI).
* Subjects who have used any drugs or substances known to be strong inhibitors or strong inducers of CYP 3A4/5 enzymes (also known as cytochrome P-450 enzymes) or P-Glycoprotein (Pgp) within 30 days prior to Period 1, Day -1. Subjects must agree to abstain from grapefruit/grapefruit juice and seville oranges for 2 days before period Ia, Day -1 and throughout the study.
* Use of other investigational drugs at the time of enrollment (consenting), or 5 half-lives of enrollment whichever is longer; or longer if required by local regulations, and for any other limitation of participation in an investigational trial based on local regulations.
* History of unstable psychiatric illness requiring medications or hospitalization within the previous 12 months.
* History of concurrent illness that required hospitalization within 14 days prior to Day 1 of the study.
* Any condition that in the clinical judgment of the Investigator would make the subject unsuitable for participation.
* Allergies or allergic reactions to any of the products used in this study.
* Subjects who have had a clinically significant illness within 4 weeks prior to Day -1.
* Subjects with QTcB interval duration >430 msec (males) or >450 (females) obtained from the ECG recorder's measurements on the screening ECG taken after at least 5 minutes of quiet rest in supine position.
* History or current evidence of clinically significant hepatic, renal, cardiovascular (i.e., deep venous thrombosis, pulmonary embolism), psychological, pulmonary, metabolic, endocrine, neurologic (i.e., transient ischemic attack or stroke within the past 6 months) infectious, gastrointestinal (i.e., any condition which may affect drug absorption) hematologic, oncologic disease, retinopathy, or other medical disorders, as determined by screening history, physical examination, laboratory test results, or 12-lead ECG.
* History of unexplained syncope.
* Subjects with creatinine clearance < 80 mL/min (based on Cockcroft-Gault equation).
* Subjects who, in the opinion of the Investigator, should not participate in the study.
* Any employee of the Duke Clinical Research Unit (DCRU).
* Subjects who have blood relatives of another study participant.
* Subjects must be compliant and meet all inclusion and exclusion criteria unless, following discussions between the Principal Investigator or his designate, it is determined that a minor exception is not indicative of clinically significant safety risk and unlikely to confound the results of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
The release profile of Ondansetron Pulsatile Release (Ond-PR) in the human gastrointestinal (GI) tract matches the one predicted from test tube dissolution experiments. | The time to reach peak blood concentration (tmax) for oral Ondansetron Standard (Ond-St) is ~2 hours (h). Therefore, tmax for Ond-PR with in vitro dissolution time of 3 - 4 h is expected to be 5 - 6 h (i.e., 3 - 4 h delay + normal absorption time).
  Serum levels of ondansetron after oral administration of Ond-PR in healthy human volunteers. Standard PK parameters will be calculated based on the serum levels to verify that the drug levels reach the peak blood concentration 5 - 6 hours after oral administration.
  Time Frame: Blood samples will be taken immediately before oral Ond-PR administration, followed by sampling at 0.5, 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6 and 10 hours after drug administration.

SECONDARY OUTCOMES:
To determine drug-drug interactions of Ond-PR with a simultaneously-administered MPh-IR. | 5 - 6 h
  For our secondary objective we plan to determine drug-drug interactions between Ond-PR and MPh-IR when they are simultaneously administered orally. Specific parameters to be assessed include changes in the PK, properties (see above for the specific parameter list), safety/tolerability profiles of Ond-PR.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Noveck, MD, PhD, Principal Investigator — Duke University; Ashwin Patkar, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States